CLINICAL TRIAL: NCT02514109
Title: Clinical, Electrophysiological and Biological Diagnostic Criteria of Sensory Neuronopathies
Status: Terminated | Type: Observational
Why Stopped: Start of a new study concerning the same patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0908074; 2009-A00679-48 (Other: ANSM)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Neuronopathy
Keywords: neuronopathy; antibodies; Clinical and biological diagnostic criteria
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for antibodies measure
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient: Male or female patient aged 18 years or more with a clinically pure sensory neuropathy, abnormal ENMG in sensory nerves in more than one limb and complete etiological assessment allowing a diagnosis of sensory neuronopathy.
  Interventions: Other: Neurological assessment and Blood sample
- control: Male or female patient aged 18 years or more with a clinically pure sensory neuropathy, abnormal ENMG in sensory nerves in more than one limb and complete etiological assessment allowing a diagnosis of sensory neuropathy excluding a neuronopathy.
  Interventions: Other: Neurological assessment and Blood sample

INTERVENTIONS:
Other: Neurological assessment and Blood sample — Neurological assessment (physical examination, electroneuromyography , International Prognostic Score (ISS), Overall Disability Scale (ODS)) and 2 blood collection tubes for antibody screening

SUMMARY:
The diagnosis of sensory neuronopathy is difficult to establish because the only certainty criterion is based on the detection of specific lesions in the posterior spinal ganglion which is usually not possible. There is to date no clinical and electrophysiological criteria or validated biomarker for the diagnosis of this type of neuropathy. In a retrospective study, we analyzed the files of patients with peripheral sensory neuronopathy certain and established clinical and electrophysiological diagnostic criteria for sensitive neuronopathy. We therefore wish now validate these criteria and investigate possible associated antibodies on a prospective cohort of patients.

DETAILED DESCRIPTION:
All the patients (patient group and control) will be included in the study after giving their consent. The clinical, biological and electrophysiological data concerning the neuropathy will be collected. There is no specific follow-up for the study.

Blood samples will be retrospectively analyzed for antibody screening.

ELIGIBILITY:
Inclusion Criteria:

* A :Patients Male or female patient aged 18 years or more with a clinically pure sensory neuropathy, abnormal ENMG in sensory nerves in more than one limb and complete etiological assessment allowing a diagnosis of sensory neuronopathy.

B :Controls Male or female patient aged 18 years or more with a clinically pure sensory neuropathy, abnormal ENMG in sensory nerves in more than one limb and complete etiological assessment allowing a diagnosis of sensory neuropathy excluding a neuronopathy.

Exclusion Criteria:

* Patient with a sensory-motor neuropathy or incomplete clinical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient group : patient with sensitive neuronopathy Control group :patient without sensitive neuronopathy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Likelihood ratio diagnostic criteria established on the study population | baseline
  The set of diagnostic criteria giving the best sensitivity and specificity for a diagnosis of sensory neuronopathy (composite measure)

SECONDARY OUTCOMES:
Identified antibodies | baseline
  Sensibility and specificity of identified antibodies (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ANTOINE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (12):
- France (12):
  - CHU Angers, Angers
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - Hopital Pitie Salpetriere, Paris
  - CHU Poitiers, Poitiers
  - Chu Saint-Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Chu de Tours, Tours